CLINICAL TRIAL: NCT05914545
Title: A PhaseⅠStudy to Evaluate the Safety, Tolerability, Pharmacokinetics and Efficacy of FZ-AD004 in Patients With Advanced Solid Tumors
Brief Title: A Study of FZ-AD004 in Patients With Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Shanghai Fudan-Zhangjiang Bio-Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: F0040-101
Record Dates: First submitted 2023-05-09; First posted 2023-06-22 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Advanced and Metastatic Solid Tumor
Keywords: Advanced and Metastatic Solid Tumor
MeSH Terms: conditions — Neoplasm Metastasis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental: FZ-AD004 (Experimental): Participants enrolled in the dose escalation part or dose expansion part
  Interventions: Drug: FZ-AD004

INTERVENTIONS:
Drug: FZ-AD004 — Dose Escalation：Subjects will receive an intravenous infusion of FZ-AD004 in a dose escalation until confirmed progression, unaccepted toxicity, or any criterion for withdrawal from the study.
  Dose Expansion：Subject will receive a single dose of FZ-AD004 at 1-2 dose level on Day1 of each cycles.
  Other Names: FZ-AD004-Antibody-drug Conjugate

SUMMARY:
This study is one single group of participants with advanced solid tumors. It is the first time the drug has been used in humans. There will be two parts including Dose Escalation and Dose Expansion to evaluate the safety, tolerability, pharmacokinetics, and clinical activity of FZ-AD004.

DETAILED DESCRIPTION:
This is a first-in-human (FIH), Phase 1, open-label, dose escalation and dose expansion study to evaluate the safety, tolerability, pharmacokinetics and preliminary efficacy of FZ-AD004 in patients with advanced/metastatic solid tumors. FZ-AD004 is administered via intravenous infusion using an accelerated titration method followed by a conventional 3 + 3 study design to identify the maximum tolerated dose (MTD) and dose-limiting toxicities（DLT）during cycle 1. In addition, the maximum-tolerated dose and recommended Phase II dose for FZ-AD004 will be determined.

ELIGIBILITY:
Inclusion Criteria:

1. Patients able to give written informed consent;
2. Age ≥ 18 and ≤ 75 years old, male or female;
3. Patients have histological or cytological diagnosis with advanced solid tumors.
4. Have measurable lesions defined in RECIST v. 1.1;
5. Expected survival ≥ 12 weeks;
6. Eastern Cancer Cooperative Group (ECOG) performance status 0-1;
7. Patients of child bearing potential must agree to take contraception during the study and for 6 months after the last day of treatment.

Exclusion Criteria:

1. Have had other malignant tumors in the past 5 years;
2. Have CNS (central nervous system) metastasis with clinical symptoms;
3. Had undergone major surgery or severe trauma within 4 weeks prior to the first dose;
4. Had undergone systemic high-dose steroids within 2 weeks of initiation of study treatment;
5. Have history of psychotropic drug abuse, alcohol or drug abuse；
6. Women who are pregnant or lactating；
7. Other circumstances that is deemed not appropriate for the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 121 (Estimated)
Dates: Start 2023-06-12 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
The dose limiting toxicity ( DLT) | 21 Days (first cycle)
  To determine the dose limiting toxicities (DLTs) of FZ-AD004.
Maximum Tolerable Dose (MTD) | 21 Days (first cycle)
  To determine the maximum tolerated dose (MTD) and/or recommended doses for expansion (RDEs). RDEs will not exceed MTD.
Adverse Events | Screening up to study completion
  To check the numbers of AEs happened during the course of trial.
Objective Response Rate (ORR) according to RECIST 1.1 | From subject randomization up to 60 months.
  To evaluate the objective response rate (ORR) [Complete Response (CR) + Partial Response (PR)] of FZ-AD004 when administered intravenously (IV) as monotherapy at the RDEs to patients with metastatic or locally advanced unresectable tumors.

SECONDARY OUTCOMES:
Progression free survival(PFS) according to RECIST 1.1 | From subject randomization up to 60 months.
  Progression-free survival (PFS) was defined as the interval from the first dose start date to the date of disease progression defined as documented progressive disease (PD) or death from any cause, whichever occurs first.
Duration of Response(DOR) according to RECIST 1.1 | From subject randomization up to 60 months
  Duration of Response was defined as the duration of overall response measured from the time measurement criteria are met for CR or PR (whichever is first recorded) until the first date that recurrent or progressive disease is objectively documented (taking as reference for progressive disease the smallest measurements recorded since the treatment started).
Overall Survival (OS) according to RECIST 1.1 | From subject randomization up to 60 months.
  Overall survival was defined as the time from the date of the first dose start date to the date of death due to any cause.
Terminal elimination half-life (t1/2) of Total Antibody, Free DXd and FZ-AD004 | Up to 17 weeks
  To check how much time Total Antibody, Free DXd and FZ-AD004 will take to eliminate half of it's concentration from participants.
Maximum observed plasma concentration (Cmax) of Total Antibody, Free DXd and FZ-AD004 | Up to 17 weeks
  o check what will be the maximum concentration participants will obtained of Total Antibody, Free DXd and FZ-AD004 in their blood plasma.
Area under the concentration-time curve (AUC 0-∞) from time 0 to infinity of Total Antibody, Free DXd and FZ-AD004 | Up to 17 weeks
  To check the drug profile for absorption, distribution, metabolism and excretion for Total Antibody, Free DXd and FZ-AD004 in participants blood plasma
Time to Cmax (Tmax) of Total Antibody, Free DXd and FZ-AD004 | Up to 17 weeks
  To check what time will it take to reach the maximum contraction of Total Antibody, Free DXd and FZ-AD004 in study participants
Number of subjects who develop detectable anti-drug antibodies (ADAs) | From subject randomization up to 60 months.
  To check the" Anti Drug Antibody" develops in participants against the FZ-AD004 through blood sample

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Chest Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: No